CLINICAL TRIAL: NCT01143103
Title: Comparison Between Respiratory Physiotherapy With Cough Assist Technique and Usual Respiratory Care in Intensive Care Patients Suffering of Neurologic Disorder
Brief Title: Comparison Between Respiratory Therapy With Cough Assist Technique and Usual Respiratory Therapy in Intensive Care Patients Suffering of Neurologic Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Didier Tassaux, MD, Intensive care unit, university hospital of Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: cough assist; cough assist (Other: University hospital of Geneva)
Record Dates: First submitted 2010-06-02; First posted 2010-06-14 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2010-06

CONDITIONS: Neurologic Disorder
Keywords: Respiratory therapy in neurologic disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Respiratory therapy with cough assist (Experimental)
  Interventions: Device: Cough assist (Philips,respironics)
- Usual respiratory therapy (Active Comparator)
  Interventions: Other: Usual respiratory therapy

INTERVENTIONS:
Device: Cough assist (Philips,respironics)
  Arms: Respiratory therapy with cough assist
Other: Usual respiratory therapy
  Arms: Usual respiratory therapy

SUMMARY:
The present study aims to compare the efficiency of respiratory therapy with cough assist and the efficiency of usual respiratory therapy in intensive care patients suffering of neurologic disorder and cough ineffectiveness. The investigators hypothesis is that cough assist is more efficient than usual respiratory care in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Peak flow < 270 ml if the patient has one of the following diagnostic: post neurosurgery status, cerebral trauma, tetraparesia or tetraplegia

Exclusion Criteria:

* Death expected in the following 24h
* Bulbar dysfunction if extubated
* pneumothorax
* intracerebral mass effect
* elevated intracranial pressure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Duration of stay in intensive care unit
Number of additional unplanned respiratory therapy treatment

SECONDARY OUTCOMES:
Duration of stay in the hospital
Pulmonary infection
Oxygenation parameters before and after respiratory therapy
Intracranial pressure elevation during respiratory therapy if an intracerebral pressure monitoring is available
Need of reintubation in the 48h following successful intubation

CONTACTS AND LOCATIONS:
Overall Officials: Didier Tassaux, Study Director — University Hospital, Geneva; Lise Piquilloud, Principal Investigator — University Hospital, Geneva
Locations (1):
- University hospital of Geneva, Geneva, Switzerland